CLINICAL TRIAL: NCT02999555
Title: Presence and Quantification of Inflammatory Cytokines, Dendritic Cells, Vasorin and Soluble Flt1 in Aspirated Follicular Fluid
Brief Title: Novel Evaluation of Aspirated Follicular Fluid
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Meir Medical Center (Other)
Collaborators: Weizmann Institute of Science (Other)
Responsible Party: Principal Investigator, Anat Hershko Klement, Dr Anat Hershko Klement, Meir Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: MMC160192-16CTIL
Record Dates: First submitted 2016-12-18; First posted 2016-12-21 (Estimated); Last update posted 2017-08-11 (Actual); Status verified 2017-08

CONDITIONS: Ovary Inflammation
MeSH Terms: conditions — Oophoritis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Aspirated follicular fluid (Experimental): Follicular fluid aspirated by follicle size and tested for the novel markers after eggs were identified and separated for the purpose of fertilization
  Interventions: Procedure: Ovum pickup

INTERVENTIONS:
Procedure: Ovum pickup — Ovum pickup or Egg retrieval, that is performed not for the purpose of the study, but for the purpose of well known in vitro fertilization indications
  Other Names: Egg retrieval

SUMMARY:
A molecular study of follicular fluid aspirated from ovarian follicles during routine in vitro fertilization treatment, after the eggs were identified and separated.

DETAILED DESCRIPTION:
Ovarian stimulation is a routine part of in vitro fertilization treatment: this process involves an inflammatory response in the developing follicles. We still do not completely understand the complex interactions leading to the maturation of the egg and the multiple interactions of the egg with its supporting cells. In this study we will assess follicular fluid, letf over after the eggs were identified and separated, for the presence of inflammatory mediators, dendritic cells , vasorin and soluble Flt1. The presence and quantification of these factors, as well as their correlation with the size of the aspirated follicle is the focus of this study.

ELIGIBILITY:
Inclusion Criteria:

* All women going through a fertility/ fertility preservation indicated egg retrieval in the in vitro fertilization (IVF) unit in 'Meir medical center',
* Patients' informed consent

Exclusion Criteria:

* Patients refusing to take part in the study

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 100 (Estimated)
Dates: Start 2017-02-01 (Actual); Primary Completion 2017-12 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
Soluble Vasorin levels | 24 hours post egg retrieval
Soluble Flt 1 levels | 24 hours post egg retrieval
Dendritic cells quantification | 24 hours post egg retrieval

CONTACTS AND LOCATIONS:
Overall Officials: MEIR medical center REB committee REB committee, Study Chair — Tel Aviv University
Locations (1):
- Meir Medical Center, Kfar Saba, Israel

REFERENCES:
- [Background] Wulff C, Wiegand SJ, Saunders PT, Scobie GA, Fraser HM. Angiogenesis during follicular development in the primate and its inhibition by treatment with truncated Flt-1-Fc (vascular endothelial growth factor Trap(A40)). Endocrinology. 2001 Jul;142(7):3244-54. doi: 10.1210/endo.142.7.8258. PMID 11416048
- [Background] Gruemmer R, Motejlek K, Berghaus D, Weich HA, Neulen J. Regulation of soluble vascular endothelial growth factor receptor (sFlt-1/sVEGFR-1) expression and release in endothelial cells by human follicular fluid and granulosa cells. Reprod Biol Endocrinol. 2005 Oct 25;3:57. doi: 10.1186/1477-7827-3-57. PMID 16248895